CLINICAL TRIAL: NCT00821288
Title: Post-treatment Care of Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Susan G. Komen Breast Cancer Foundation (Other)
Responsible Party: Principal Investigator, Dawn L. Hershman, Associate Professor of Medicine & Epidemiology, Columbia University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: AAAC5741; DISP0706868 (Other Grant/Funding Number: The Susan Komen Foundation)
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Breast Neoplasm
Keywords: cancer survivorship; survivorship prescription; cancer related anxiety
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Survivorship Intervention (Experimental): Latina and Caucasian breast cancer survivors treated in an urban academic medical center receiving Survivorship Intervention
  Interventions: Behavioral: Survivorship Intervention
- Facing Forward (Active Comparator): Latina and Caucasian breast cancer survivors treated in an urban academic medical center receiving Survivorship Intervention Facing Forward: Life after Cancer Treatment manual
  Interventions: Behavioral: Facing Forward

INTERVENTIONS:
Behavioral: Survivorship Intervention — Survivorship Consultation is a one hour consultation in a survivorship clinic. The consultation will be performed by a nurse practitioner under the supervision of a medical oncologist. The consultation will result in a detailed written document outlining the individuals "Survivorship Prescription" including treatment summary, surveillance recommendations, risk for late-effects, cancer screening recommendations, genetic risk, and life style recommendations. This written document will be provided to the patient and her treating physician. In addition, referrals will be made to appropriate adjunct services as needed (e.g. psychologist, nutritionist, social worker).
  Other Names: Survivorship Prescription
  Arms: Survivorship Intervention
Behavioral: Facing Forward — Facing Forward: Life after Cancer Treatment is a guide for people who were treated for cancer published by the NCI. It is a 24-page manual that summarized many key issues of interest to cancer survivors during the re-entry phase, and contains sections on medical care after treatment, symptoms after treatment, feelings after treatment, social relationships after cancer treatment, and dealing with practical matters such as insurance and employment. The manual is available in English and Spanish. This will be given at the time of registration and the table of contents will be reviewed with the patient.
  Other Names: Life after Cancer Treatment manual
  Arms: Facing Forward

SUMMARY:
The overall goal of this proposal is to improve the post-treatment care of breast cancer survivors and to understand the barriers to optimal post-treatment care in Latina and Non-Hispanic women.

DETAILED DESCRIPTION:
The proposed investigation is a randomized prospective evaluation of a Survivorship Intervention in improving the quality of care, treatment satisfaction and understanding of care in Latina and Caucasian breast cancer survivors treated in an urban academic medical center. Patients will be recruited within 6 weeks of completing their last definitive breast cancer therapy (radiation or chemotherapy). Patients will complete self administered baseline and follow-up questionnaires. Following baseline evaluation patients will be randomized to receiving either written information for follow-up care of cancer survivors published by the National Cancer Institute (Facing Forward), or the Survivorship Intervention. Patients will not be aware that they are participating in a randomized intervention. After verbally agreeing to participate they will be randomized to group A or B and will receive the corresponding consent. Patients will be re-assessed 3 and 6 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be screened for the following inclusion criteria:
* Age >18 years
* History of stage 0, I, II, or IIIa breast cancer and no evidence of recurrent disease
* Within 6 weeks of completion of breast cancer therapy (Surgery, Radiation or Chemotherapy)
* Caucasian and/or Hispanic (English or Spanish-speaking)
* Willing to undergo a 1 hr cancer survivorship evaluation

Exclusion Criteria:

* Patients with the following active conditions or behaviors will be excluded from participation:
* Evidence of recurrent or metastatic breast cancer
* Patients who have received surgery only with no adjuvant therapy
* Uncontrolled or significant psychiatric illness/social situations that would preclude completion of questionnaire or follow-up evaluation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in FACIT-TS questionnaire score | Baseline, 6 months
  This is designed to measure change in positive health related behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn L Hershman, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia Unviersity Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hershman DL, Greenlee H, Awad D, Kalinsky K, Maurer M, Kranwinkel G, Brafman L, Jayasena R, Tsai WY, Neugut AI, Crew KD. Randomized controlled trial of a clinic-based survivorship intervention following adjuvant therapy in breast cancer survivors. Breast Cancer Res Treat. 2013 Apr;138(3):795-806. doi: 10.1007/s10549-013-2486-1. Epub 2013 Mar 31. PMID 23542954